CLINICAL TRIAL: NCT03574428
Title: A Randomised, Double-Blind, Placebo Controlled, Single Ascending Doses Study With GNbAC1 in Healthy Male Volunteers
Brief Title: Single Ascending Doses Study With GNbAC1 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeNeuro Australia PTY Ltd (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-006
Record Dates: First submitted 2018-05-16; First posted 2018-07-02 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Active Comparator): GNbAC1 36 mg/kg single i.v. dose or GNbAC1 placebo
  Interventions: Drug: GNbAC1; Other: GNbAC1 Placebo
- Cohort 2 (Active Comparator): GNbAC1 60 mg/kg single i.v. dose or GNbAC1 placebo
  Interventions: Drug: GNbAC1; Other: GNbAC1 Placebo
- Cohort 3 (Active Comparator): GNbAC1 85 mg/kg single i.v. dose or GNbAC1 placebo
  Interventions: Drug: GNbAC1; Other: GNbAC1 Placebo
- Cohort 4 (Active Comparator): GNbAC1 110 mg/kg single i.v. dose or GNbAC1 placebo
  Interventions: Drug: GNbAC1; Other: GNbAC1 Placebo

INTERVENTIONS:
Drug: GNbAC1 — Monoclonal Antibody infused i.v.
Other: GNbAC1 Placebo — Equivalent to GNbAC1 Buffer

SUMMARY:
This is a phase I, double-blind, placebo controlled, parallel group, dose-escalating, randomised study designed to assess and compare the safety and tolerability, PK, and immunogenicity of GNbAC1 administered as a single dose at 4 different dose levels of 36, 60, 85 and 110 mg/kg.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy male volunteers
* Negative urine drug screen
* Have signed the informed consent.

Main Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Use of any prescription medication within 30 days prior to the administration of investigational product and/or non-prescription medication (including herbal and natural remedies, homeopathy, vitamins, and minerals) within 7 days prior to the administration of investigational product or anticipated use of any concomitant medication during the study. Permissible exceptions are paracetamol up to 4g/day ceasing a minimum of 12 hours prior to infusion and Ibuprofen up to 1.2g/day ceasing a minimum of 24 hours prior to infusion. Paracetamol and ibuprofen are allowed during the study, but only 24 hours after completion of the administration of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses of GNbAC1 (Serious Adverse Events, Adverse Events) | 57 days
  Serious Adverse Events (SAE), Adverse Events (AE)

SECONDARY OUTCOMES:
Pharmacokinetic (PK): GNbAC1 serum concentrations over time | 57 days
  GNbAC1 serum concentrations over time
Immunogenicity: Antibodies against GNbAC1 (ADA) | 57 days
  Antibodies against GNbAC1 (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research Ltd, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Porchet H, Vidal V, Kornmann G, Malpass S, Curtin F. A High-dose Pharmacokinetic Study of a New IgG4 Monoclonal Antibody Temelimab/GNbAC1 Antagonist of an Endogenous Retroviral Protein pHERV-W Env. Clin Ther. 2019 Sep;41(9):1737-1746. doi: 10.1016/j.clinthera.2019.05.020. Epub 2019 Jul 13. PMID 31311668